CLINICAL TRIAL: NCT06555588
Title: Engage: A Randomized Controlled Trial Testing the Efficacy of a Telehealth-Delivered Psychosocial Intervention to Decrease Symptom Interference in Patients With Advanced Cancer
Brief Title: Engage Psychosocial Intervention for Cancer Symptoms
Acronym: Engage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00115646; R01CA291768 (NIH)
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Advanced Breast Cancer; Advanced Prostate Cancer; Advanced Lung Cancer; Advanced Colorectal Carcinoma; Advanced Colorectal Adenocarcinoma
Keywords: Acceptance and Commitment Therapy; Cognitive Behavioral Therapy; Pain management; Fatigue management; Symptom management; Telehealth; Psychosocial intervention
MeSH Terms: conditions — Agnosia | interventions — engage 8200; Palliative Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned with equal (1:1) allocation to either ENGAGE or Supportive Care. A stratified block randomization scheme will be used to ensure group balance based on: 1) the primary outcome of symptom interference (i.e., less than 7 vs. 7 to 10); and 2) cancer type (i.e., breast, prostate, lung, or colorectal).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENGAGE (Experimental): Behavioral symptom management focused on values identification and skills training.
  Interventions: Behavioral: ENGAGE
- Supportive Care (Active Comparator): Education, support, and resources focused on common cancer-related concerns.
  Interventions: Behavioral: Supportive Care

INTERVENTIONS:
Behavioral: ENGAGE — This intervention is delivered by trained therapists over four, 45-60 minute, manualized telehealth sessions. The session content is based on an integration of Cognitive Behavioral Therapy (CBT) and Acceptance and Commitment Therapy (ACT) approaches for managing symptoms of pain, fatigue, and distress. Participants are trained in behavioral symptom management skills (e.g., activity pacing, mindfulness) with an emphasis on engaging in highly valued activities.
  Arms: ENGAGE
Behavioral: Supportive Care — This intervention is delivered by trained therapists over four, 45-60 minute, manualized telehealth sessions. The session content is designed to provide participants with education, support, and resources for a range of issues relevant to those with advanced cancer (e.g., education on symptoms, body image concerns, and financial concerns).
  Arms: Supportive Care

SUMMARY:
The goal of this clinical trial is to test the efficacy a new psychosocial symptom management intervention called ENGAGE for patients with Stage IV breast, prostate, lung, or colorectal cancer. Participants will be randomized to ENGAGE or a Supportive Care intervention. Patient-reported outcomes will be assessed at baseline, 2 months, and 4 months.

DETAILED DESCRIPTION:
Pain, fatigue, and distress are highly prevalent, co-occurring, and interfering symptoms in patients with advanced cancer. This trial will test a brief telehealth delivered psychosocial intervention called ENGAGE. ENGAGE aims to help patients decrease symptom interference and improve their quality of life. Patients with Stage IV cancer (breast, prostate, lung, or colorectal) and moderate-to-severe symptom interference will be randomized to ENGAGE or Supportive Care. Patient-reported outcomes will be assessed at baseline, 2 months, and 4 months. Aim 1 is to determine ENGAGE's efficacy for reducing symptom interference (primary outcome) at 2 months (primary endpoint). Aim 2 is to determine ENGAGE's efficacy for improving secondary outcomes at 2 months. Aim 3 is to test the maintenance of ENGAGE's effects on primary and secondary outcomes at 4 months. An exploratory aim seeks insights for future implementation efforts using mixed-methods data collection from patients, oncology providers, and clinic leaders.

ELIGIBILITY:
Inclusion Criteria:

* Receiving cancer care at a Duke Cancer Network (DCN) clinic
* Oncologist confirmed Stage IV breast, prostate, lung, or colorectal cancer
* Worst pain, fatigue, or distress rated at >/= 3 out of 10 in the past 7 days for at least 2 symptoms
* MD Anderson Symptom Inventory (MDASI) Interference with Daily Living Scale average score of >/= 3 out of 10 in the past 7 days
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or lower
* At least 18 years old
* Ability to speak and read English
* Hearing and vision that allows for successful completion of telehealth sessions

Exclusion Criteria:

* Significant cognitive impairment indicated in medical chart or during telephone screening on a mental status questionnaire
* Serious psychiatric condition (e.g., schizophrenia, suicidal intent) that would contraindicate safe study participation
* Participation in the last 6 months in Cognitive-Behavioral Therapy or Acceptance and Commitment Therapy for cancer symptom management
* Enrollment in hospice at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
MD Anderson Symptom Inventory (MDASI) Interference with Daily Living Scale | 2 months
  This measure assesses the degree to which, over the past 7 days, symptoms of pain, fatigue, and/or distress have interfered with patients' general activity, mood, work (including work around the house), relations with other people, walking, and enjoyment of life. Items are scored from 0 = "Did not interfere" to 10 = "Interfered completely," and averaged for a composite score.

SECONDARY OUTCOMES:
MD Anderson Symptom Inventory (MDASI) Interference with Daily Living Scale | 4 months
  This measure assesses the degree to which, over the past 7 days, symptoms of pain, fatigue, and/or distress have interfered with patients' general activity, mood, work (including work around the house), relations with other people, walking, and enjoyment of life. Items are scored from 0 = "Did not interfere" to 10 = "Interfered completely," and averaged for a composite score.
MD Anderson Symptom Inventory (MDASI) Symptom Severity Scale | 2 months and 4 months
  This measure assesses the severity of pain, fatigue, and distress at their worst over the past 7 days. Items are scored from 0 = "not present" to 10 = "as bad as you can imagine". Each item is interpreted individually, with higher scores reflecting worse symptom severity.
Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Symptoms | 2 months and 4 months
  This measure assesses patients' level of confidence to manage or control their symptoms, manage their symptoms in different settings, and to keep symptoms from interfering with work, relationships, or personal care. Items are scored from 1 = "I am not confident at all" to 5 = "I am very confident." Items are summed and converted to T-scores, with higher scores indicating better self-efficacy.
Openness to Experience subscale of the Comprehensive Assessment of Acceptance and Commitment Therapy (CompACT) | 2 months and 4 months
  This subscale assesses patients' openness to experience difficult thoughts, emotions, and sensations (i.e., psychological acceptance). Items are scored from 0 = "strongly disagree" to 6 = "strongly agree," with higher scores indicating more acceptance. Items are averaged for a composite score.
Behavioral Awareness subscale of the Comprehensive Assessment of Acceptance and Commitment Therapy (CompACT) | 2 months and 4 months
  This subscale assesses patients' level of present moment awareness (i.e., mindfulness). Items are scored from 0 = "strongly disagree" to 6 = "strongly agree," with higher scores indicating more mindfulness. items are averaged for a composite score.
Valued Action subscale of the Comprehensive Assessment of Acceptance and Commitment Therapy (CompACT) | 2 months and 4 months
  This subscale assesses patients' degree of values identification and willingness to take actions that align with their personal values. Items are scored from 0 = "strongly disagree" to 6 = "strongly agree," with higher scores indicating more values identification and engagement. Items are averaged for a composite score.
Brief Pain Inventory (BPI) | 2 months and 4 months
  This pain severity measure assesses pain at its worst, least, average, and now. Response options range from 0 = "no pain" to 10 = "pain as bad as you can imagine". items are averaged for a composite score.
Brief Fatigue Inventory (BFI) | 2 months and 4 months
  This fatigue severity measure assesses fatigue over the last 7 days from 0 = "no fatigue" to 10 = "as bad as you can imagine" at its usual, worst, and right now. Items are averaged for a composite score.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety-Short Form | 2 months and 4 months
  This anxiety symptom measure assesses fear, worry, uneasiness, nervousness, and tension. Response options range from 1 = "never" to 5 = "always." Items are summed and converted to T-scores, with higher scores indicating worse anxiety symptoms.
Patient-Reported Outcomes Measurement Information System (PROMIS) Depression-Short Form | 2 months and 4 months
  This depressive symptoms measure assesses worthlessness, helplessness, hopelessness, depressed mood, failure, and sadness. Response options range from 1 = "never" to 5 = "always." Items are summed and converted to T-scores, with higher scores indicating worse depressive symptoms.
Functional Assessment of Cancer Therapy-General (FACT-G) | 2 months and 4 months
  This quality of life measure is composed of 4 subscales: physical, social/family, emotional, and functional well-being. Items are rated on a 0 = "not at all" to 4 = "very much" scale and summed for subscale scores and an overall quality of life score.
Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp) | 2 months and 4 months
  This measure includes an overall spiritual well-being score and three subscales: 1) meaning (i.e., reason for living, sense of meaning and purpose); 2) peace (i.e., feeling peaceful, sense of harmony within oneself); and 3) faith (i.e., finding strength and comfort in faith or spiritual beliefs). Response options range from 0 = "not at all" to 4 = "very much"; two items are reverse coded. Higher scores indicate greater spiritual well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Cancer Network, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of this trial will be presented at professional meetings and published in peer-reviewed journals. The dataset will be made available to qualified investigators within 6 months of the publication of the primary outcome paper. The dataset will contain necessary identifiers, excluding those prohibited by HIPAA. The investigators will be required to sign a data use agreement and obtain Institutional Review Board (IRB) approval before receiving the data set.
  Public use study data and associated documentation will also be made available to the research community through the National Cancer Institute's Cancer Data Service (CDS) data repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The dataset will be made available to qualified investigators within 6 months of the publication of the primary outcome paper. Data will be available for at least 6 years.
Access Criteria: The dataset and supporting information will be made available to qualified investigators to allow replication of analyses or secondary data analyses. The PI will review requests for data access. The investigators will be required to sign a data use agreement and obtain IRB approval before receiving the data set. The mechanism for data sharing will be reviewed by the IRB. The investigators requesting the data will need to cite the original study.
  Users of the public use data must register with National Cancer Institute's Cancer Data Service (CDS) and agree to the Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity. Data users also agree not to share or redistribute any data downloads.

REFERENCES:
- [Derived] Winger JG, Kelleher SA, Yu JA, Ma JE, Majestic CM, Martinson EB, Olsen MK, Lerebours R, Sutton LM, Somers TJ. Engage: Protocol of a randomized controlled trial of a telehealth-delivered psychosocial intervention to decrease symptom interference in patients with advanced cancer. Contemp Clin Trials. 2025 Sep;156:108053. doi: 10.1016/j.cct.2025.108053. Epub 2025 Aug 18. PMID 40834926